CLINICAL TRIAL: NCT03127709
Title: A Clinical, Structural, and Functional Neuroimaging Study of Cognition in Adults With Erdheim-Chester Disease, Langerhans Cell Histiocytosis, Rosai-Dorfman Disease, and Other Histiocytoses
Brief Title: A Study of Memory, Thinking, and Brain Imaging in Adults With Histiocytosis
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 17-199
Record Dates: First submitted 2017-04-11; First posted 2017-04-25 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Histiocytosis
Keywords: 17-199; histiocytosis
MeSH Terms: conditions — Histiocytosis | interventions — Trail Making Test; Wechsler Scales; Neuropsychological Tests; 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Participants with a histiocytic disorder diagnosis: Participants will have a histiocytic disorder as determined by a corroborating constellation of histopathology, clinical, and/or radiologic findings.
  Interventions: Behavioral: Trail Making Test, Parts A & B; Behavioral: Brief Test of Attention; Behavioral: Symbol Span; Behavioral: Controlled Oral Word Association Test; Behavioral: The Hopkins Verbal Learning Test-Revised; Behavioral: Brief Visuospatial Memory Test-Revised; Behavioral: Hospital Anxiety and Depression Scale; Behavioral: McGill Quality of Life Scale; Diagnostic Test: MR Brain Imaging; Diagnostic Test: Resting state functional MRI; Behavioral: Functional Assessment of Cancer Therapy Cognitive Scale (FACT-Cog)

INTERVENTIONS:
Behavioral: Trail Making Test, Parts A & B — Part A is a timed measure of visual scanning and graphomotor speed. Part B is a timed measure of cognitive flexibility.
Behavioral: Brief Test of Attention — Assesses auditory working memory
  Other Names: BTA
Behavioral: Symbol Span — Assesses visual working memory
  Other Names: WMS-IV
Behavioral: Controlled Oral Word Association Test — The COWA timed test of phonemic verbal fluency. It requires the subject to generate as many words as possible, beginning with a given letter of the alphabet (i.e., F, A, and S).
  Other Names: COWA
Behavioral: The Hopkins Verbal Learning Test-Revised — HVLT-R is a test of verbal learning and memory. Scores obtained are the total number of words.
  Other Names: HVLT-R
Behavioral: Brief Visuospatial Memory Test-Revised — The BVMT-R is a test of visuospatial learning and memory.
  Other Names: BVMT-R
Behavioral: Hospital Anxiety and Depression Scale — The HADS is a brief assessment validated in many cancer populations.
  Other Names: HADS
Behavioral: McGill Quality of Life Scale — This is a questionnaire that is a validated 17-item QOL instrument validated for ill patients and in the particular context of the ancer.
  Other Names: McGill QOL
Diagnostic Test: MR Brain Imaging — Standard of care brain MR imaging includes high-resolution 3D T1-weighted images in the axial plane. The axial T1-weighted images will be isotropic with a typical matrix size of 256 x 256, 256 mm field-of-view (FOV) and 1 mm slice thickness covering the whole brain.
Diagnostic Test: Resting state functional MRI — Scanning will be performed on a 3 Tesla General Electric scanner (Optima 750W) with a GEM HNU 24-channel head coil. rsFMRI matching the FLAIR and T1 post-contrast images will be obtained. For resting state fMRI, T2*-weighted images will be acquired with a single-shot gradient echo echo-planar imaging (EPI) sequence in the axial orientation (TR = 2500 ms, TE = 30 ms, FA = 80°, slice thickness = 4 mm, FOV= 240mm2, matrix=64×64) covering whole brain. For the resting state fMRI portion of the scan, patients will be instructed by the technologist or research staff to leave eyes open, focus on looking at a crosshair, and not think about anything during the scan.
  Other Names: rsFMRI
Behavioral: Functional Assessment of Cancer Therapy Cognitive Scale (FACT-Cog) — This is a validated 37-item QOL instrument for cancer patients with cognitive complaints. The measures consist of FACT-Cog total, perceived cognitive impairments, perceived cognitive abilities, and impact on quality of life.

SUMMARY:
The purpose of this study is to try to understand how histopcytosis can cause symptoms or problems in the brain. The tests being done in the study will look at memory and thinking as well as brain function via MRI scan.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years.
* Fluency in English
* Diagnosis of a histiocytic disorder as determined, in the opinion of the study PI, by a corroborating constellation of histopathology, clinical, and/or radiologic findings.
* Will undergo Standard of Care MRI.

Exclusion Criteria:

* Known intracranial involvement of histiocytosis (including dura, leptomeninges and brain parenchyma)
* Prior stroke or intracranial hemorrhage
* Other (non-histiocytic) intracranial neoplasm or neurological disorder deemed by the PI or Co-PI to confound neuroimaging studies (e.g., demyelinating disease)
* Existing diagnosis of a psychiatric disorder or untreated mood disturbance
* Existing diagnosis of a neurodegenerative disease, such as Alzheimer's disease
* Chronic or daily excessive alcohol consumption as determined by the PI.
* History of chronic use of corticosteroids, defined as continuous treatment for six months or longer at any time in the past
* History of severe claustrophobia or other contraindications to patient SOC brain MRI
* Prior intravenous cytarabine or cladribine
* Other current or prior treatments (e.g., high-dose chemotherapy for a different cancer) deemed by the PI or Co-PI to confound imaging studies or cognitive performance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will have a diagnosis of a histiocytic disorder as determined, in the opinion of the study PI, by a corroborating constellation of histopathology, clinical, and/or radiologic findings.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
neurocognitive function | 1 year
  Neurocognitive tests will yield raw scores that are converted to z-scores, normalized for participant's age, sex and educational level.The proportion of participants demonstrating cognitive impairment (as defined by 2 or more z-scores less than -1.5) will be summarized. Also, the proportion of participants with impairment (z < -1.5) for each cognitive test will be summarized. In this way the cognitive assessment yields a dichotomous outcome of impaired versus not impaired for each participant but also allow for more granular assessment of impairment in specific cognitive domains.
quality of life | 1 year
  questionnaires will yield raw scores (total score for HADS and McGill QOL, as well as anxiety and depression subscores for the HADS). QOL scores will be analyzed as raw scores. Cognitive test scores will be transformed into z-sores (based on score distributions from established normative samples with a mean of 0 and standard deviation of 1) to define the presence/severity of cognitive dysfunction. Scores will be normalized for age, sex and education.
comparing of grey matter volume | 1 year
  In a whole-brain analysis, first, cortical thickness will be compared between participants and controls and regions of statistically significant grey matter loss will be identified. This is done computionally with a whole-brain, vertex-by-vertex approach, as stated above. Also, as stated above (Section 7), statistical significance thresholding is at p<0.001, correcting for multiple comparisons using the False Discovery Rate (FDR) method and clustering thresholds, methods used in various high-throughput contexts, including MRI analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Eli Diamond, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering — http://mskcc.org